CLINICAL TRIAL: NCT00492908
Title: Randomized Clinical Trial Comparing A Titanium-Nitride-Oxide Coated Stent With A Zotarolimus-Eluting Stent in Patients With Coronary Artery Disease
Brief Title: Randomized Trial Comparing Titan Stent With Zotarolimus-Eluting Stent
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Department of Cardiology, Bern University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KEK237_06
Record Dates: First submitted 2007-06-25; First posted 2007-06-27 (Estimated); Last update posted 2014-05-01 (Estimated); Status verified 2014-04

CONDITIONS: Coronary Heart Disease
Keywords: Coronary Revascularization; Titanium-Nitride-Oxide Coated Stent; Zotarolimus-Eluting Stent
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Titanium Nitride Oxide Coated Stent (Active Comparator): Stent
  Interventions: Device: Helistent Titan2 (Titanium coated stent)
- Zotarohlimus Eluting Stent (Active Comparator): Stent
  Interventions: Device: EndeavorTM (Zotarolimus-Eluting Stent)

INTERVENTIONS:
Device: Helistent Titan2 (Titanium coated stent) — Titan2
  Arms: Titanium Nitride Oxide Coated Stent
Device: EndeavorTM (Zotarolimus-Eluting Stent) — Endeavor
  Arms: Zotarohlimus Eluting Stent

SUMMARY:
A Randomized Comparison of a Titanium-Nitride-Oxide Coated Stent (Helistent Titan2, Hexacath) With a Zotarolimus-Eluting Stent (EndeavorTm, Medtronic) for Percutaneous Coronary Intervention

DETAILED DESCRIPTION:
Objectives: The purpose of this study is to compare the Titanium-Nitride-Oxide Coated Stent (Helistent Titan2, Hexacath) with a Zotarolimus-Eluting Stent (EndeavorTm, Medtronic) in a non-inferiority trial.

Design: Prospective, multi-center, randomized, non-inferiority trial to be conducted at 3 Swiss interventional cardiology centers. Patients will be randomized in a single-blind fashion (1:1 randomization) to either the Titanium-Nitride-Oxide Coated Stent (Helistent Titan2, Hexacath) or the Zotarolimus-Eluting Stent (EndeavorTm, Medtronic).

Study Population: Patients with symptomatic coronary artery disease including patients with chronic stable angina, silent ischemia, unstable angina, and non-ST elevation myocardial infarction, who qualify for percutaneous coronary interventions

Antiplatelet Therapy: Aspirin 100 mg qd indefinitely; Clopidogrel 75 mg qd for 3 months

Enrollment: A total of 300 patients will be enrolled

All patients will undergo repeat angiography at 6-8 months.

All patients will be followed for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

The following patients are eligible for inclusion

1. Age ≥18 years
2. Symptomatic coronary artery disease including patients with chronic stable angina, silent ischemia, unstable angina, and non-ST elevation myocardial infarction
3. Presence of one or more coronary artery stenoses >50% in a native coronary artery from 2.25 to 4.0 mm in diameter that can be covered with one or multiple stents;
4. No limitation on the number of treated lesions, and vessels, and lesion length

Exclusion Criteria:

1. Pregnancy
2. Known intolerance to aspirin, clopidogrel, heparin, stainless steel, titan, zotarolimus or contrast material
3. Inability to provide informed consent
4. Currently participating in another trial before reaching first endpoint
5. ST segment elevation myocardial infarction (STEMI)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2007-06; Primary Completion 2009-03 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
In-stent late luminal loss | 6-8 months after stent implantation

SECONDARY OUTCOMES:
TLR, TVR, Death or MI, CV death or MI, CV death, Death, MI, Stent thrombosis, Stenosis, Restenosis | 30 days, 6-8 months, 1, 2, 3, 4 and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Windecker, MD, Principal Investigator — Department of Cardiology, University Hospital Bern, Bern, Switzerland
Locations (1):
- Department of Cardiology, University Hospital Bern, Bern, Switzerland

REFERENCES:
- [Background] Windecker S, Simon R, Lins M, Klauss V, Eberli FR, Roffi M, Pedrazzini G, Moccetti T, Wenaweser P, Togni M, Tuller D, Zbinden R, Seiler C, Mehilli J, Kastrati A, Meier B, Hess OM. Randomized comparison of a titanium-nitride-oxide-coated stent with a stainless steel stent for coronary revascularization: the TiNOX trial. Circulation. 2005 May 24;111(20):2617-22. doi: 10.1161/CIRCULATIONAHA.104.486647. Epub 2005 May 9. PMID 15883209
- [Background] Windecker S, Mayer I, De Pasquale G, Maier W, Dirsch O, De Groot P, Wu YP, Noll G, Leskosek B, Meier B, Hess OM; Working Group on Novel Surface Coating of Biomedical Devices (SCOL). Stent coating with titanium-nitride-oxide for reduction of neointimal hyperplasia. Circulation. 2001 Aug 21;104(8):928-33. doi: 10.1161/hc3401.093146. PMID 11514381
- [Derived] Pilgrim T, Raber L, Limacher A, Wenaweser P, Cook S, Stauffer JC, Garachemani A, Moschovitis A, Meier B, Juni P, Windecker S. Five-year results of a randomised comparison of titanium-nitride-oxide-coated stents with zotarolimus-eluting stents for coronary revascularisation. EuroIntervention. 2015 Mar;10(11):1284-7. doi: 10.4244/EIJY15M01_04. PMID 25572026
- [Derived] Pilgrim T, Raber L, Limacher A, Loffel L, Wenaweser P, Cook S, Stauffer JC, Togni M, Vogel R, Garachemani A, Moschovitis A, Khattab AA, Seiler C, Meier B, Juni P, Windecker S. Comparison of titanium-nitride-oxide-coated stents with zotarolimus-eluting stents for coronary revascularization a randomized controlled trial. JACC Cardiovasc Interv. 2011 Jun;4(6):672-82. doi: 10.1016/j.jcin.2011.02.017. PMID 21700254